CLINICAL TRIAL: NCT05106712
Title: Effects of Vitamin D Supplementation on Reproductive, Hormonal and Metabolic Profiles, and on IVF Outcomes, in PCOS Infertile Saudi Women : a Randomized-controlled Clinical Trial
Brief Title: Vitamin D Supplementation and Improvement of PCOS Therapy and IVF Outcomes in Infertile Saudi Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Ramya Sindi, Assistant Professor in Assisted Reproduction Technology, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (AMSEC 82/1-4-2021)
Record Dates: First submitted 2021-10-08; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Female Infertility; Polycystic Ovary Syndrome; Pathologic Processes; Vitamin D Deficiency; IVF; Vitamin D Supplement
Keywords: Polycystic Ovary Syndrome; IVF; Vitamin D; Randomized Clinical Trial
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome; Pathologic Processes; Vitamin D Deficiency | interventions — Cholecalciferol; Clomiphene; Letrozole

STUDY DESIGN:
Intervention Model Description: the present intervention trial is designed to achieve the following two objectives: 1) measurement of the therapeutic effects of Vitamin D3 supplement alone and in combination with an ovulation-inducing agent (e.g., Clomiphene citrate or Letrozole) on the ovarian functional status and the hormonal and metabolic features of PCOS-Vitamin D-deficient infertile Saudi women; and 2) measurement of the effectiveness of Vitamin D3 supplement versus placebo on the clinical pregnancy rate, fertilization implantation rate, live birth rate, and other outcome parameters following in-vitro fertilization (IVF) application in PCOS-Vitamin D-deficient infertile patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and most researchers will be unaware of the actual grouping. Only two investigators who will be not involved in participant management or data analysis will be aware of the grouping. Vitamin D3, Clomiphene citrate, Letrozole and placebo pills with identical package, size, color and appearance will be used in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D3 (Experimental): Participants will be treated with oral vitamin D3 4000IU capsules per day for around 12 weeks
  Interventions: Drug: Vitamin D3
- Ovulation-inducing drug "Clomiphene citrate" (Active Comparator): Participants will be treated with oral Clomiphene citrate using its respective "Stair-step dosage protocol" as follow: 50 mg, 100 mg, and 150 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively.
  Interventions: Drug: Clomiphene Citrate
- Ovulation-inducing drug "Letrozole" (Active Comparator): Participants will be treated with oral Letrozole using its respective "Stair-step dosage protocol" as follow: 5 mg, 5 mg, and 7.5 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively, respectively.
  Interventions: Drug: Letrozole
- Placebo (Placebo Comparator): PCOS-Vitamin D-deficient infertile women in the control (Placebo) group will be treated with equal amount of placebo tablets per day for the same duration.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Vitamin D3 — 4000IU per day for around 12 weeks.
  Arms: Vitamin D3
Drug: Clomiphene Citrate — oral Clomiphene citrate using its respective "Stair-step dosage protocol" as follow: 50 mg, 100 mg, and 150 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively.
  Arms: Ovulation-inducing drug "Clomiphene citrate"
Drug: Letrozole — oral Letrozole using its respective "Stair-step dosage protocol" as follow: 5 mg, 5 mg, and 7.5 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively, respectively.
  Arms: Ovulation-inducing drug "Letrozole"
Other: placebo — participants in the control (Placebo) group will be treated with equal amount of placebo tablets per day for the same duration
  Arms: Placebo

SUMMARY:
This randomized double-blinded-controlled clinical trial consists of two protocols as follow: protocol 1: evaluation of the therapeutic effects of Vitamin D3 supplement when given alone and in combination with an ovulation-inducing agent (e.g., Clomiphene citrate or Letrozole) on ovarian functional status and hormonal and metabolic features of PCOS-Vitamin D-deficient infertile Saudi women; and protocol 2: evaluation of the effectiveness of Vitamin D3 supplement versus placebo on the clinical pregnancy rate, fertilization implantation rate, live birth rate, and other outcome parameters following in-vitro fertilization (IVF) application in these PCOS-Vitamin D-deficient infertile patients.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is one of the most common endocrinological and metabolic disorders that affect women at their reproductive age and leading to female infertility worldwide. PCOS exhibits multiple etio-pathogenic properties in which the genetic, nutritional, behavioral and environmental factors are intertwined to its complexity and heterogeneity. At that respect, impaired vitamin D status (hypo-vitaminosis D) has recently gained an immense interest as a leading cause in development of PCOS and the prevalence of its underlying hormonal/metabolic abnormalities and ovarian malfunctions. Additionally, serum levels of vitamin D are considered as potential predictors of successful Assisted Reproductive technology (ART) outcomes in infertile women with PCOS or with unexplained infertility. Most importantly, it is hypothesized that vitamin D supplementation improve the hormonal and metabolic profile and reproduction activity in treatment naïve PCOS and vitamin D deficient patient women; and also improve the pregnancy rate and oocyte and embryos' quality following in vitro fertilization (IVF) in these PCOS-vitamin D deficient infertile women. In despite, evidence regarding the therapeutic value of vitamin D supplementation for treatment of PCOS and improving IVF outcomes in PCOS-vitamin D-deficient infertile Saudi women population remain scarce. Therefore, the present study is designed to achieve the following two objectives: 1) measurement of the therapeutic effects of Vitamin D3 supplement alone and in combination with an ovulation-inducing agent (e.g., Clomiphene citrate or Letrozole) on the ovarian functional status and the hormonal and metabolic features of PCOS-Vitamin D-deficient infertile Saudi women; and 2) measurement of the effectiveness of Vitamin D3 supplement versus placebo on the clinical pregnancy rate, fertilization implantation rate, live birth rate, and other outcome parameters following in-vitro fertilization (IVF) application in PCOS-Vitamin D-deficient infertile patients.

To achieve the 1st objective, the investigators plan to recruit about 450 eligible patients accounting for 10% loss to follow-up and regard a significance level at 0.05 and a power of 80%. The eligible participants will be randomized into 5 groups (1:1:1:1:1) to receive the following therapies: Group 1: monotherapy with oral vitamin D3 capsules (4000IU/day) for around 12 weeks; Group 2: monotherapy with oral Clomiphene citrate pills using its respective standard Stair-Step Dosage protocol (i.e., 50 mg, 100 mg, and 150 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively); Group 3: monotherapy with oral Letrozole pills using its respective standard Stair-Step Dosage protocol (i.e., 2.5 mg, 5 mg, and 7.5 mg, once daily for 5 days, in the 1st, 2nd, and 3rd cycle, respectively); Group 4: dual therapy with Vitamin D3 plus Clomiphene citrate by using their above mentioned dosage regimen; and Group 5: dual therapy with Vitamin D3 plus Letrozole by using their above mentioned dosage regimen. At the end of the intervention protocol, post-treatment improvements in menstrual regularity, ovulation induction rate, and ovarian volumes will be considered as the primary outcome measures, while the baseline (weak 0) and post-treatment (WK12) levels of fasting plasma glucose levels, insulin resistance (IR) indices, and serum levels of 25(OH)D, calcium, sex-hormones, reproductive mediators and adipocytokines, and lipid profile levels will be measured in the different groups and used as the secondary outcomes measures.

To achieve the 2nd objective, the investigators plan to recruit about 180 eligible PCOS-vitamin D-deficient infertile women scheduled for IVF accounting for 10% loss to follow-up and regard 0.05 significance level and 80% power. The eligible participants will be randomized into 2 groups (1:1) to receive daily oral capsules of 4000IU vitamin D3 (Group 1) or placebo (Group 2) for around 12 weeks until the day of triggering. All IVF procedures will be carried out according to the routine methods applied in ART centers. The primary outcome measures will include post-IVF clinical pregnancy, fertilization implantation, and live birth rates in both groups. Post-treatment changes in insulin resistance indices and serum levels of 25(OH)D, calcium, sex-hormones, reproductive mediators and adipocytokines, and lipid profile levels will also be measured as the secondary outcomes measures.

In both protocols, the diagnosis of PCOS is according to the revised Rotterdam PCOS consensus criteria as the presence of at least 2 of the following 3 diagnostic criteria: oligo- and(or) anovulation defined as a history of delayed menstrual cycle >35 days in length or ≤9 spontaneous bleeding episodes per year, clinical and(or) biochemical evidence of hyperandrogenism, and features of polycystic ovaries detected by ultrasound (≥12 follicles of 2-9 mm in size found in at least one ovary and/or having ovarian volume more than 10 cm3). The eligible infertile women will be considered "treatment naïve PCOS" if they have PCOS and they had no taken any prior anti-PCOS medication; and they will be considered "vitamin D deficient" if they have fasting serum 25(OH)D ≤20 ng/mL according to The Endocrine Society Clinical Practice Guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20 to 42 years old;
2. Diagnosed with PCOS (Rotterdam Criteria);
3. Written informed consent.

Exclusion Criteria:

1. Non-PCOS Infertile patients, e.g, who have Cushing's syndrome, congenital adrenal hyperplasia, androgen-secreting tumors, hyperprolactinemia.
2. PCOS patients who are underwent any anti-infertility treatments.
3. PCOS patients who had receiving any vitamin D supplement or any multivitamin supplement within the past 3 month prior to enrollment process.
4. PCOS patients with established diagnosis of diabetes mellitus, chronic liver, kidney, or thyroid diseases.
5. PCOS patients receiving any treatment affect the metabolism of vitamin D.
6. Any supplements that contain vitamin D within the past month.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile Saudi women
Enrollment: 700 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Clinical pregnancy | through study completion, an average of 18 months
  Clinical pregnancy is defined as at least one gestational sac on ultrasound at around 7 weeks' gestation with the detection of heart beat activity after the completion of the first embryo transfer
Number of Participants with live birth | through study completion, an average of 18 months
  Live birth is defined as the delivery of at least one baby after 24 weeks of gestation that exhibits any sign of life

SECONDARY OUTCOMES:
Number of participants with Pregnancy loss rate | through study completion, an average of 18 months
  Pregnancies that result in a abortion at any point throughout pregnancy
Number of participants with improved metabolic parameters | through study completion, an average of 18 months
  Pre- and post-intervention plasma levels of glucose, insulin, vitamin D, reproductive adipocytokines, and lipid profile